CLINICAL TRIAL: NCT05940753
Title: Flashmobstudie Landelijke Meting Reisbereidheid Medisch Oncologische Zorg
Brief Title: Flash Mob Study With Regard to Travel Willingness Among Patients With Cancer
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 15954
Record Dates: First submitted 2023-03-20; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Cancer
Keywords: oncology; hospital choice; willingness to travel
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: medical oncology patients in the out-patient clinic or treatment unit on 13 or 14 march 2023: No interventions.
  Interventions: Other: Survey about travel willingness regarding cancer treatment and follow-up

INTERVENTIONS:
Other: Survey about travel willingness regarding cancer treatment and follow-up — No intervention. Willingness to travel is examined through a survey. The survey will be conducted digitally, but may also be done on paper. In the survey a minimal set of categorized patient data (e.g. age, gender, level of education) is collected as part of the survey. For patients who cannot independently complete the questionnaire (for example due to low literacy skills), a volunteer, medical student or researcher is allowed to help the patient.

SUMMARY:
This is a cross-sectional study in the form of a flash mob study, in which an inventory will be made on 13 and 14 March 2023 of the willingness to travel of oncology patients in the participating hospitals. Patients who have an appointment with an internist-oncologist or oncology specialist nurse at the outpatient clinic or by telephone and patients who come to day treatment unit for medical oncology are asked to participate. Willingness to travel is examined by means of a survey, in which a minimal set of categorized patient data (e.g. age, gender, level of education) is collected as part of the survey.

ELIGIBILITY:
Inclusion criteria:

* Medical oncology patients with an appointment in the out-patient clinic or day treatment unit on 13 or 14 march 2023
* Medical oncology patients with an (video) call appointment in the out-patient clinic on 13 or 14 march 2023

Exclusion criteria:

* Patients in the inpatients oncology unit
* Medical oncology patients with no appointment on 13 or 14 march 2023

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical Oncology patients who have an (call) appointment with our medical oncology outpatient clinic and/or day treatment unit on 13 or 14 march 2023.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Travel willingness | 1 day
  How far is the oncological patient willing to travel for his/her systemic treatment or follow-up?

SECONDARY OUTCOMES:
Facilitating and inhibiting factors for willingness to travel | 1 day
  What are facilitating and inhibiting factors in patients' willingness to travel?
Which patient characteristics are associated with willingness to travel? | 1 day
  Which patient characteristics are associated with willingness to travel? (age, type of cancer, curative/palliative treatment, distance to nearest hospital)

CONTACTS AND LOCATIONS:
Overall Officials: An KL Reyners, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided